CLINICAL TRIAL: NCT02965001
Title: Phase II Trial: uPAR-PET/CT for Prognostication in Head- and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Louise Madeleine Risør, Principal investigator, medical doctor, Ph.D student, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 366_16
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Head and Neck Cancer
Keywords: Molecular Imaging; uPAR-PET/CT; Head and neck cancer; curative intended radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-NOTA-AE105 (Experimental): All participants have an uPAR-PET/CT scan performed before initiation of the routine radiotherapy
  Interventions: Drug: 68Ga-NOTA-AE105

INTERVENTIONS:
Drug: 68Ga-NOTA-AE105 — The patients are refered to an uPAR-PET/CT scan before initiation of the routine radiotherapy and the prognostic efficacy is assessed by registration of recurrence rate and death at routine clinical follow-up.
  Other Names: uPAR

SUMMARY:
Head and neck cancer (HNC) is the 6th most common cancer worldwide. In the last decade, there has been made substantial improvements in diagnosis, staging and treatment of HNC. The overall survival has improved, but for some subgroups it is unchanged and therefore new prognostic and surveillance methods are warranted.

One of the hallmarks in cancer is the ability to invade the surrounding tissue and metastasize. Studies have shown that the urokinase proteolytic plasminogen activator (uPA) and its receptor (uPAR) are present at the very front of the invasive tumor and they are considered essential in cancer invasion and metastasis. Consequently, an uPAR-targeted tracer offers a very promising target for functional PET imaging and may be a stronger prognostic marker compared to routine FDG-PET/CT. We wish to clarify how uPAR-PET/CT correlate to patient outcome compared to routine FDG-PET/CT in patients with HNC in the pharynx, larynx and oral cavity, who are referred to curative intended radiotherapy. In this project all participants have an uPAR-PET/CT scan performed before initiation of the routine radiotherapy and the prognostic efficacy is determined by assessment of the recurrence rate and mortality at routine clinical follow-up.

DETAILED DESCRIPTION:
In this study all included patients with head and neck cancer (HNC) have an uPAR-PET/CT scan performed before the initiation of the curative intended radiotherapy. After the radiotherapy treatment the patients attend the routine clinical follow-up programme at Rigshospitalet to follow the loco-regional control, signs of metastasis and the overall survival. These relapse- and survival parameters will be correlated to the SUVmax, SUVmean and the TNM stage obtained from the uPAR scan and will be compared to the findings on the routine FDG scan to clarify which tracer is the strongest prognostic marker in HNC.

If any previous tissue samples have been taken from the tumour before the patient enters the study the uPAR immunohistopathology of the tissue sample will be compared to the uPAR-PET/CT findings. We will not perform any biopsies or tissue samples in this study.

ELIGIBILITY:
Inclusion Criteria:The patient

* has a diagnosis of biopsy-verified cancer of the pharynx, larynx or oral cavity
* is referred to curative intended radiotherapy
* understands the given information and has given informed consent and
* age above 18 years.

Exclusion Criteria:

Pregnancy, lactation/breast feeding, age above 85 years, obesity (bodyweight above 140 kg), small cancers of the larynx (1A,1B), allergy to 68Ga-NOTA-AE105, metastasis on FDG-PET/CT, other previously known cancers, claustrophobia.

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Freedom from any failure | 1-3 years

SECONDARY OUTCOMES:
Overall Survival | 1-3 years
Disease free survival | 1-3 years
Distant metastasis free survival | 1-3 years
Loco-regional control | 1-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kjær, Professor, Study Director — Rigshospitalet, Denmark
Locations (1):
- Departmen of Physiology, Nuclear Medicine and PET, Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Risor LM, Clausen MM, Ujmajuridze Z, Farhadi M, Andersen KF, Loft A, Friborg J, Kjaer A. Prognostic Value of Urokinase-Type Plasminogen Activator Receptor PET/CT in Head and Neck Squamous Cell Carcinomas and Comparison with 18F-FDG PET/CT: A Single-Center Prospective Study. J Nucl Med. 2022 Aug;63(8):1169-1176. doi: 10.2967/jnumed.121.262866. Epub 2021 Dec 2. PMID 34857658